CLINICAL TRIAL: NCT02315885
Title: Biomarkers to Measure Treatment Response for Alcohol Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Chamindi Seneviratne, MD, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HP-00060091
Record Dates: First submitted 2014-12-05; First posted 2014-12-12 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Alcohol Dependence
Keywords: healthy volunteers; social drinkers; alcohol
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo alcohol (Placebo Comparator): <0.05% alcohol
  Interventions: Other: Alcohol administration; Placebo administration
- alcohol middle dose (Active Comparator): alcohol dose=0.45g/kg for women and 0.5g/kg for men
  Interventions: Other: Alcohol administration; Placebo administration
- alcohol high dose (Active Comparator): alcohol dose=0.90g/kg for women and 1.0g/kg for men
  Interventions: Other: Alcohol administration; Placebo administration

INTERVENTIONS:
Other: Alcohol administration; Placebo administration — consumption of 3 alcohol doses (2 regular and one placebo) each within 2h on separate days

SUMMARY:
The purpose of the research study of the K23 award is to develop a blood test that can check how much alcohol a person has consumed in the past few days. We will enroll heavy social drinkers who do not have alcohol-related problems but used to drinking 5 or more beers on a single occasion. Both men and women between ages 21 and 65 years can join the study. All participants must be of European decent.

ELIGIBILITY:
Inclusion Criteria:

* Experienced binge drinking episode(s) (5 or more standard drinks for men and 4 or more standard drinks for women consumed in about 2 hours according to NIAAA definition) in the past 30 days

Exclusion Criteria:

* DSM-IV diagnosed alcohol dependence, other drug dependencies including nicotine dependence

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-07; Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Validity of using serotonin transporter mRNA expression levels | Within 24 hours of blood sample collection and in archived blood samples from the same participant stores at -80 degrees celsius for a duration of 6 months or more from the collection date
  Validity of using serotonin transporter mRNA expression levels in 5 HTTLPR:LL and rs 25531:AA genotype carriers, as a biomarker of alcohol consumption levels.

CONTACTS AND LOCATIONS:
Overall Officials: Chamindi Seneviratne, Principal Investigator — csenevi@som.umaryland.edu
Locations (1):
- Clinical Neurobehavioral Center, Columbia, Maryland, United States